CLINICAL TRIAL: NCT06693752
Title: Pilot Study of Improved Diagnosis and Monitoring of Hydrocephalus in Neonates and Infants Using Contrast-Enhanced Ultrasound
Brief Title: CEUS Evaluation of Hydrocephalus in Neonates and Infants
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Misun Hwang, MD, Sponsor Investigator, Children's Hospital of Philadelphia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24-022232
Record Dates: First submitted 2024-11-11; First posted 2024-11-18 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Hydrocephalus in Infants; Hydrocephalus Acquired
Keywords: Ultrasound; Contrast-enhanced ultrasound; Infant hydrocephalus
MeSH Terms: interventions — Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Brain contrast-enhanced ultrasound (Experimental): The study duration per subject will be up to 30 minutes including the time to prepare the contrast agent, perform the pre-contrast imaging and the contrast-enhanced ultrasound (CEUS), as well as the 60-minute monitoring period after the administration of the contrast agent. A second CEUS exam may be performed within 1-2 weeks from the first scan for up to two CEUS exams of 1 hour and 30-minute duration each. Study participation will be complete when the 60-minute monitoring period of the last CEUS performed is complete.
  Interventions: Drug: Sulfur Hexafluoride Lipid Type A Microspheres 25 mg Injection Powder for Suspension [LUMASON]

INTERVENTIONS:
Drug: Sulfur Hexafluoride Lipid Type A Microspheres 25 mg Injection Powder for Suspension [LUMASON] — Injection of Sulfur hexafluoride lipid-type A microspheres contrast agent will be performed via the existing peripheral intravenous line using the FDA-recommended dose of 0.03 mg/kg before performing the contrast-enhanced ultrasound. The weight-based dose of 0.03 mL per kg will be repeated one time during a single examination. Following each injection, an intravenous flush of 0.9% Sodium Chloride is injected.

SUMMARY:
Hydrocephalus affects up to 2 out of every 500 births and results in long-term disability in up to 78% of those affected. The standard treatment of hydrocephalus is cerebrospinal fluid (CSF) diversion via placement of an invasive ventricular shunt to relieve elevated intracranial pressure (ICP). The clinical decision for CSF diversion is based on the ventricular size and clinical symptoms which are not robust indicators of brain health in neonatal hydrocephalus. The purpose of this study is to assess the safety and feasibility of performing brain contrast-enhanced ultrasound (CEUS) in neonates and infants with diagnosed and/or suspected hydrocephalus.

DETAILED DESCRIPTION:
Contrast-enhanced ultrasound (CEUS) is a clinically used imaging technique that uses gas-filled microbubbles to enhance the visualization of blood vessels. Ultrasound contrast agents have been approved for use in Europe for around two decades, and in the United States, the FDA has approved the use of Lumason, a second-generation lipid/sulfur hexafluoride ultrasound contrast agent, for the evaluation of focal hepatic lesions, opacification of the left ventricular chamber of the heart and assessment of vesicoureteral reflux in pediatric patients. Unlike computed tomography or magnetic resonance imaging (MRI) contrast agents, ultrasound contrast agents have no associated renal toxicity and do not require ionizing radiation or sedation. The risk of adverse events is the lowest of all contrast agents available, with only minor adverse events reported in children, such as altered taste, tinnitus, light-headedness, and nausea.

Previous investigation on cerebral physiology in hydrocephalus has shown that increasing ventricular dilation results in reduced cerebral blood flow, as well as reduced cerebral oxygen saturation and higher oxygen extraction. These findings have been studied with currently available tools such as transcranial Doppler, MRI, and near infrared spectroscopy (NIRS).

However, there is no standardized tool for robust assessment of brain health in neonatal hydrocephalus. In this regard, prior work by the study team has shown a promising brain CEUS biomarker of ICP and brain ischemia in the porcine neonatal hydrocephalus model. Specifically, cerebral microvascular flows as measured using brain CEUS correlated with invasively measured ICP and brain ischemia. Therefore, there is a dire need to introduce better imaging tools such as CEUS to the clinical setting that can detect changes in ICP and brain ischemia in patients with hydrocephalus at an early stage and prompt therapeutic implementation/monitoring. The study seeks to validate first the safety and feasibility of performing brain CEUS in neonatal hydrocephalus.

Injection of Lumason contrast agent will be performed via the existing peripheral intravenous line or central line using the FDA-recommended dose of up to 0.03 mg/kg. Contrast-agent injection will be performed twice per CEUS scan to ensure image quality and test reproducibility. Two bolus injections will performed to evaluate for dynamic brain perfusion and several 2-minute cine clips as well as static images will be acquired during the exam.

Baseline and demographic characteristics will be summarized by standard descriptive statistics. Qualitative analysis will be performed by visual rating by 2 teams, blinded to clinical information, consisting of primary investigator and second radiologist (co-investigator). Each scan will be rated for diagnostic quality and qualitative rating of cranial perfusion. Quantitative analysis will be performed using time-intensity based analysis and the particle image and/or tracking velocimetry (PIV/PTV) method. These calculations will be performed after transferring the DICOM data obtained during the research procedure. The purpose is to utilize post-processing techniques available to the study team.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females younger than 1.5 years old with diagnosed and/or suspected hydrocephalus.
2. Post menstrual age of 26 weeks or older.
3. Inpatients at the Children's Hospital of Philadelphia.
4. Parental/Legally authorized representative permission.

Exclusion Criteria:

1. Medical history of Lumason hypersensitivity.
2. Hemodynamic instability as defined by rapid escalation of cardiopulmonary support in the past 12-24 hours, as defined by the clinical care team.
3. Respiratory instability as defined by rapid escalation of respiratory support in the past 12-24 hours (Increased fraction of inspired oxygen (FiO2) requirement and/or nitric oxide).

Ages: 1 Minute to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of brain contrast-enhanced ultrasound (CEUS) examinations in infants with hydrocephalus | Up to 2 years
  Total number and percentage of successfully competed brain CEUS with adequate quality. Sufficient quality to be interpreted by radiologists without significant motion degradation and/or obscuration due to poor acoustic penetration. Visual rating by 2 teams consisting of primary investigator and second radiologist (co-investigator). Each scan will be rated for diagnostic quality and qualitative rating of cranial perfusion. The visual rating scale used will be: 0 (absent flow), 1 (decreased flow), 2 (normal flow), 3 (increased flow).
Safety of brain contrast-enhanced ultrasound (CEUS) examinations in infants with hydrocephalus | Up to 2 years
  Total number/percentage of patients who experienced adverse events (if any) will be reported to assess safety. All subjects entered into the study and receiving at least one injection of investigational drug will be included in the safety analysis. Adverse events will be recorded at 1) 60 minutes post-scanning when the monitoring period is completed, and 2) through 48 hours post-scanning, with documentation at 48 hours post-scanning if no adverse event presents until this point.

SECONDARY OUTCOMES:
Correlation between contrast-enhanced ultrasound (CEUS) parameters (intensity perfusion) and invasively measured intracranial pressure (ICP) in infants with hydrocephalus | Up to 2 years
  Pearson's or Spearman's correlation coefficients will be calculated to measure the relationship between CEUS parameters and ICP measurements. The investigators will analyze blood flow intensity perfusion as the first CEUS parameter. The correlation values will range from -1 to +1, where positive values indicate measurements increase together, negative values indicate one increases as the other decreases, and values closer to ±0.5 suggest strong relationships. The choice between Pearson's or Spearman's correlation will depend on whether the data follows a normal distribution pattern.
Correlation between contrast-enhanced ultrasound (CEUS) parameters (particle-tracking velocimetry) and invasively measured intracranial pressure (ICP) in infants with hydrocephalus | Up to 2 years
  Pearson's or Spearman's correlation coefficients will be calculated to measure the relationship between CEUS parameters and ICP measurements. The investigators will analyze particle-tracking velocimetry as the second CEUS parameter. The correlation values will range from -1 to +1, where positive values indicate measurements increase together, negative values indicate one increases as the other decreases, and values closer to ±0.5 suggest strong relationships. The choice between Pearson's or Spearman's correlation will depend on whether the data follows a normal distribution pattern.
Correlation between contrast-enhanced ultrasound (CEUS) parameters (particle-image velocimetry) and invasively measured intracranial pressure (ICP) in infants with hydrocephalus | Up to 2 years
  Pearson's or Spearman's correlation coefficients will be calculated to measure the relationship between CEUS parameters and ICP measurements. The investigators will analyze particle-image velocimetry as the third CEUS parameter. The correlation values will range from -1 to +1, where positive values indicate measurements increase together, negative values indicate one increases as the other decreases, and values closer to ±0.5 suggest strong relationships. The choice between Pearson's or Spearman's correlation will depend on whether the data follows a normal distribution pattern.
Correlation between contrast-enhanced ultrasound (CEUS) parameters (intensity perfusion) and cerebral ischemia biomarkers (lactate level and lactate/pyruvate ratio in cerebrospinal fluid) in infants with hydrocephalus | Up to 2 years
  Pearson's or Spearman's correlation coefficients will be calculated to measure the relationship between CEUS parameters and blood markers that indicate brain tissue damage due to reduced blood flow (cerebral ischemia biomarkers). The investigators will analyze blood flow intensity perfusion as the first CEUS parameter. The correlation values will range from -1 to +1, where positive values indicate measurements increase together, negative values indicate one increases as the other decreases, and values closer to ±0.5 suggest strong relationships. The choice between Pearson's or Spearman's correlation will depend on whether the data follows a normal distribution pattern.
Correlation between contrast-enhanced ultrasound (CEUS) parameters (particle-tracking velocimetry) and cerebral ischemia biomarkers (lactate level and lactate/pyruvate ratio in cerebrospinal fluid) in infants with hydrocephalus | Up to 2 years
  Pearson's or Spearman's correlation coefficients will be calculated to measure the relationship between CEUS parameters and blood markers that indicate brain tissue damage due to reduced blood flow (cerebral ischemia biomarkers). The investigators will analyze particle-tracking velocimetry as the second CEUS parameter. The correlation values will range from -1 to +1, where positive values indicate measurements increase together, negative values indicate one increases as the other decreases, and values closer to ±0.5 suggest strong relationships. The choice between Pearson's or Spearman's correlation will depend on whether the data follows a normal distribution pattern.
Correlation between contrast-enhanced ultrasound (CEUS) parameters (particle-image velocimetry) and cerebral ischemia biomarkers (lactate level and lactate/pyruvate ratio in cerebrospinal fluid) in infants with hydrocephalus | Up to 2 years
  Pearson's or Spearman's correlation coefficients will be calculated to measure the relationship between CEUS parameters and blood markers that indicate brain tissue damage due to reduced blood flow (cerebral ischemia biomarkers). The investigators will analyze particle-image velocimetry as the third CEUS parameter. The correlation values will range from -1 to +1, where positive values indicate measurements increase together, negative values indicate one increases as the other decreases, and values closer to ±0.5 suggest strong relationships. The choice between Pearson's or Spearman's correlation will depend on whether the data follows a normal distribution pattern.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No